CLINICAL TRIAL: NCT06399861
Title: Humidity in Incubators for Tiny Infants (HumidITI) Trial
Brief Title: Humidity in Incubators for Tiny Infants
Acronym: HumidITI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Matthew Rysavy, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSC-MS-24-0206
Record Dates: First submitted 2024-04-26; First posted 2024-05-06 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Extremely Premature Infant
Keywords: Humidification Protocol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Incubator ambient relative humidity (RH) of 70% (Active Comparator): Infants will be provided usual delivery room care and then placed in an incubator on admission to the NICU, receiving ambient relative humidity (RH) of 70% in the incubator.
  Interventions: Device: Incubator ambient relative humidity (RH) of 70%
- Incubator ambient relative humidity (RH) of 90% (Experimental): Infants will be provided usual delivery room care and then placed in an incubator on admission to the NICU, receiving ambient relative humidity (RH) of 90% in the incubator.
  Interventions: Device: Incubator ambient relative humidity (RH) of 90%

INTERVENTIONS:
Device: Incubator ambient relative humidity (RH) of 70% — The incubator will be set to an ambient relative humidity (RH) of 70%.
  Arms: Incubator ambient relative humidity (RH) of 70%
Device: Incubator ambient relative humidity (RH) of 90% — The incubator will be set to an ambient relative humidity (RH) of 90%.
  Arms: Incubator ambient relative humidity (RH) of 90%

SUMMARY:
The objective of the study is to assess 2 different initial incubator humidification protocols for infants <25 weeks' gestation admitted to the neonatal intensive care unit (NICU). The hypothesis is that a higher starting humidity decreases dehydration and results in no difference in survival or morbidity. Higher (90%) and lower (70%) starting humidity will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Inborn infant of <25 weeks' gestation admitted to the NICU

Exclusion Criteria:

* Infants with known congenital skin conditions
* Outborn infants
* Infants with unknown gestational age prior to birth

Ages: 0 Days to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 350 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy as assessed by percent of birth weight lost | upon admission to the NICU, postnatal week 2
Composite safety score | from time of admission to the NICU through hospital discharge (about 4-5 months)
  A single composite safety score will be reported (mortality and 6 morbidities will be assessed to determine this score). The composite score ranges from 0 to 7, with a higher score indicating a better outcome, as listed below:
  * 0 = Infant does not survive
  * 1 = Infant survives, has all 6 assessed morbidities
  * 2 = Infant survives, has 5 assessed morbidities
  * 3 = Infant survives, has 4 assessed morbidities
  * 4 = Infant survives, has 3 assessed morbidities
  * 5 = Infant survives, has 2 assessed morbidities
  * 6 = Infant survives, has 1 assessed morbidities
  * 7 = Infant survives, has no assessed morbidities
  Morbidities assessed:
  * grade III-IV intraventricular hemorrhage (IVH)
  * surgical necrotizing enterocolitis (NEC) or focal intestinal perforation (FIP)
  * grade III bronchopulmonary dysplasia (BPD)
  * treated retinopathy of prematurity (ROP)
  * culture-proven late-onset sepsis (LOS)
  * patent ductus arteriosus (PDA) ligation

SECONDARY OUTCOMES:
Average axillary temperatures in degrees Celsius (°C) | from time of admission to the NICU to postnatal day 3
Average daily total fluid intake in milliliters per kilogram per day (mL/kg/d) | from time of admission to the NICU to postnatal day 14
Average daily total fluid output in milliliters per kilogram per day (mL/kg/d) | from time of admission to the NICU to postnatal day 14
Average daily weight in grams | from time of admission to the NICU to postnatal day 14
Average daily sodium administered in milliequivalents per kilogram per day (mEq/kg/d) | from time of admission to the NICU to postnatal day 14
Average daily serum sodium in milliequivalents per liter per day (mEq/L/d) | from time of admission to the NICU to postnatal day 14
Average daily calories administered in kilocalories per kilogram per day (kcal/kg/d) | from time of admission to the NICU to postnatal day 14
Average daily protein administered in grams per kilogram per day (g/kg/d) | from time of admission to the NICU to postnatal day 14
Number of participants who were administered insulin | from time of admission to the NICU to postnatal day 14
Number of participants who were administered vasopressor | from time of admission to the NICU to postnatal day 14
Weight | 36 weeks postmenstrual age
Length | 36 weeks postmenstrual age
Head circumference | 36 weeks postmenstrual age
Number of participants who survive to hospital discharge | from time of admission to the NICU to discharge (about 4-5 months)
Number of participants with severe (grade III-IV) intraventricular hemorrhage (IVH) | from time of admission to the NICU to discharge (about 4-5 months)
Number of participants with necrotizing enterocolitis (NEC) or focal intestinal perforation (FIP) | from time of admission to the NICU to discharge (about 4-5 months)
Number of participants with grade III bronchopulmonary dysplasia (BPD) | from time of admission to the NICU to discharge (about 4-5 months)
Number of participants with treated retinopathy of prematurity [ROP] | from time of admission to the NICU to discharge (about 4-5 months)
Number of participants with culture-proven late-onset sepsis (LOS) | from time of admission to the NICU to discharge (about 4-5 months)
Number of participants with patent ductus arteriosus (PDA) ligation | from time of admission to the NICU to discharge (about 4-5 months)
Number of unplanned removals of vascular access or breathing tube | from time of admission to the NICU to postnatal day 14

OTHER OUTCOMES:
Average total pre-discharge costs | from time of admission to the NICU to discharge (about 4-5 months)
  Total pre-discharge costs (assessed from the health system perspective) encompass facility costs and professional service costs.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A. Rysavy, MD, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (6):
- United States (6):
  - Nationwide Children's Hospital - Grant Medical Center, Columbus, Ohio
  - Nationwide Children's Hospital - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Children's Memorial Hermann Hospital, Houston, Texas
  - The Woman's Hospital of Texas, Houston, Texas
  - St. Luke's Baptist Hospital, San Antonio, Texas
  - North Central Baptist Hospital, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No